CLINICAL TRIAL: NCT03061929
Title: Human Milk Composition in Indian Mothers
Status: Completed | Type: Observational
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Other Study IDs: AL21
Record Dates: First submitted 2017-02-09; First posted 2017-02-23 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Breast Feeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Undernourised: Mother's with BMI less than 18.5
- Normally Nourished: Mother's with BMI greater than or equal to 18.5 to less than or equal to 25.
- Overnourished: Mother's with BMI over 25 to less than or equal to 35.

SUMMARY:
Nutritional profile of mother's milk is influenced by various factors including environmental, dietary and nutritional status of the mother. Given the huge diversity noted in nutritional status and ethnic dietary patterns in Indian population, including pregnant and lactating mothers, it can be conceivably predicted to have an influence on milk composition. With the lack of recent literature addressing these, it is vital to understand and update the influence if any, of nutritional status and dietary patterns on nutritional quality of human milk. The proposed Human milk analysis clinical study in Indian mothers is aimed to achieve a more recent and updated database of nutritional profile of Indian mother's milk considering the dietary and regional influences and demographic differences which can play a key role in levels of nutrients in mother's milk. In order to incorporate the varied dietary patterns, milk samples will be collected from mothers recruited from 8 sites across the country and analysed for important nutrient levels.

DETAILED DESCRIPTION:
The study is a 5-month prospective observational cohort study. Approximately 258 mother-infant pairs in 33-42 weeks of pregnancy will be recruited. Eligibility assessment will be done for the mother at enrolment and for the mother-infant pair at delivery. Based on the recorded anthropometric data and BMI (kg/m2) calculated based on the self-reported pre-pregnancy weight or earliest recorded body weight from their first trimester, mothers consenting to the study will be categorized as either well-nourished or malnourished. All study centers will recruit equal number of participants in each group at their respective sites. As per standard of care, mothers will continue to take the prenatal supplement primarily consisting of folic acid, elemental iron, calcium and will be encouraged to breast feed their infants during prenatal visits. Breastfeeding advice normally consists of messages on the benefits of breastfeeding, instructions on early initiation of breastfeeding and proper breastfeeding techniques, and recommendation on exclusive breastfeeding for the first 6 months. Mothers will be provided with a diary to make a note about their supplement intake and the frequency of breastfeeding. The entry of the details will be enquired telephonically (biweekly) and restated during the face follow-up sessions at study visits 3 and 4.

ELIGIBILITY:
Inclusion Criteria:

1. Mother is at 33 to 42 weeks of pregnancy, is between 20 and 35 years of age and is contactable by telephone
2. Mother is non smoker and non alcoholic.
3. Mother has BMI 35 kg per m2 based on self reported pre pregnant weight or the earliest measured weight during the first trimester from the hospital record.
4. Mother confirms her intention to breast feed for 4 months.
5. Infant is a singleton with a gestational age of greater than 37 to 42 weeks and is able to feed from the mother normally.
6. Infants born between 33 to 37 weeks, by definition are preterm, but is not declared very low birth weight by the pediatrician, and is able to feed from the mother normally.
7. Infant is judged to be in good health in the opinion of the investigator.
8. Mother or Legally Acceptable Representative has voluntarily signed and dated an Informed Consent Form, approved by an Independent Ethics Committee/Institutional Review Board (IEC/IRB) or other applicable privacy regulation authorization prior to any participation in the study.

Exclusion Criteria:

1. An adverse maternal, fetal or infant medical history that is thought by the investigator to have potential effects on infant's growth and or development. This includes but is not limited to suspected maternal substance abuse such as alcohol or drug.
2. Mother has known gestational diabetes and/or a diagnosis of pre-eclampsia.
3. Mother with contraindications to breastfeeding such as known HIV or conditions that can significantly interfere with breastfeeding such as serious illness as per investigator's judgment.
4. Mother had a breast surgery.
5. Mother and or newborn infant has major illness that requires intensive care admission 24 hours.
6. Infant is advised to be kept in NICU and unable to feed from the mother for more than a week or has a medical history that is thought by the investigator to have potential effects on infant's growth and or development.
7. Infant has major congenital anomaly in the PI's opinion
8. Participation in another study that has not been approved as a concomitant study by AN.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 258 mother-infant pair subjects (86 per group) will be enrolled. The mothers will be normally-nourished or undernourished or over nourished based on pre-pregnancy measured BMI (kg/m2).
Sampling Method: Probability Sample
Enrollment: 248 (Actual)
Dates: Start 2017-03-24 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Change in fat content of milk | from 15 days post-partum to 98 days post-partum
  Fat content will be analyzed by standardized and modern analytical methods.

SECONDARY OUTCOMES:
Change in fatty acid profile in mother's milk | from 15 days post-partum to 98 days post-partum
  Fatty acid content in milk will be analyzed by standardized and modern analytical methods
Assessment of dietary intake of macro and micronutrients by mother | From 15 days post-partum to 98 days post-delivery
  Dietary intake of the mother will be assessed by a food frequency questionnaire (FFQ). Nutrient analysis of the FFQ will be done using a standardized nutrient database.

CONTACTS AND LOCATIONS:
Overall Officials: Deepti Khanna, Ph.D., Study Chair — Abbott Nutrition Research & Development
Locations (8):
- India (8):
  - MS Ramaiah Medical College and Hospital, Bangalore
  - Sir Gangaram Hospital, Delhi
  - Institute of Child Health, Kolkata
  - Institute of Post Graduate Medical Education & Research and SSKM Hospital, Kolkata
  - King George Medical College & University, Lucknow
  - Cheluvumba Hospital, Mysore
  - King Edward Memorial Hospital, Pune
  - Sant Dnyadneshwar Medical Institute, Pune

IPD SHARING:
Plan to Share IPD: No